CLINICAL TRIAL: NCT03562871
Title: An Open-label, Randomized, Phase I/II Trial Investigating the Safety and Efficacy of IO102 in Combination With Pembrolizumab, With or Without Chemotherapy, as First-line Treatment for Patients With Metastatic Non-Small Cell Lung Cancer
Brief Title: IO102 With Pembrolizumab, With or Without Chemotherapy, as First-line Treatment of Metastatic NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IO Biotech (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IO102-012 / KN-764; 2018-000139-28 (EudraCT Number); KEYNOTE-764 (Other: Merck Sharp & Dohme Corp)
Record Dates: First submitted 2018-05-14; First posted 2018-06-20 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: NSCLC
Keywords: PD-1; PD-L1; Programmed Cell Death 1; Chemotherapy; Pemetrexed; Carboplatin; Pembrolizumab; Immunotherapy; IO102; Keytruda
MeSH Terms: interventions — pembrolizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A1 (Experimental): Drug: IO102 100µg administered subcutaneously (SC) on Day 1 of each 3 week cycle PLUS Drug: pembrolizumab (Keytruda) 200 mg intravenous (IV) infusion on Day 1 of each 3 week cycle
  Interventions: Biological: IO102; Biological: pembrolizumab (Keytruda)
- Cohort A2 (Active Comparator): Drug: pembrolizumab (Keytruda) 200 mg IV infusion on Day 1 of each 3 week cycle
  Interventions: Biological: pembrolizumab (Keytruda)
- Cohort B1 (Experimental): Drug: IO102 100µg SC on Day 1 of each 3 week cycle PLUS Drug: pembrolizumab (Keytruda) 200 mg IV on Day 1 of each 3 week cycle PLUS Drug: carboplatin (Carboplatin Kabi) at a target AUC of 5 mg/mL IV infusion on Day 1 of each 3 week cycle for a max of 4 administrations PLUS Drug: pemetrexed (Pemetrexed Alvogen) at 500 mg/m2 IV infusion on Day 1 of each 3 week cycle
  Interventions: Biological: IO102; Biological: pembrolizumab (Keytruda); Drug: Carboplatin (Carboplatin Kabi); Drug: Pemetrexed (Pemetrexed Alvogen)
- Cohort B2 (Active Comparator): Drug: pembrolizumab (Keytruda) 200 mg IV on Day 1 of each 3 week cycle PLUS Drug: carboplatin (Carboplatin Kabi) at a target AUC of 5 mg/mL IV infusion on Day 1 of each 3 week cycle for a max of 4 administrations PLUS Drug: pemetrexed (Pemetrexed Alvogen) at 500 mg/m2 IV infusion on Day 1 of each 3 week cycle
  Interventions: Biological: pembrolizumab (Keytruda); Drug: Carboplatin (Carboplatin Kabi); Drug: Pemetrexed (Pemetrexed Alvogen)

INTERVENTIONS:
Biological: IO102 — test immunotherapy
  Arms: Cohort A1; Cohort B1
Biological: pembrolizumab (Keytruda) — anti-PD-1 immunotherapy
Drug: Carboplatin (Carboplatin Kabi) — chemotherapy
  Arms: Cohort B1; Cohort B2
Drug: Pemetrexed (Pemetrexed Alvogen) — chemotherapy
  Arms: Cohort B1; Cohort B2

SUMMARY:
The purpose of this study is to determine if IO102 combined with pembrolizumab with or without chemotherapy is safe tolerable and effective in the treatment of Non-small Cell Lung Carcinoma (NSCLC).

The hypothesis is that IO102 will improve the objective response rate (ORR) in patients with metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic NSCLC or non squamous NSCLC
* Have biomarker-positive solid tumor
* Male participants of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study medication through 120 days after the last dose of study medication
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication
* The participant must provide written informed consent
* Have measurable disease per RECIST 1.1
* Have provided a blood sample and archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher immune-related AE (irAE)
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Radiotherapy within 2 weeks of start of trial treatment
* Vaccination with a live vaccine within 30 days prior to the first dose of trial treatment.Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of trial treatment.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years.
* Has known active CNS metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity (≥Grade 3) to IO102, pembrolizumab, carboplatin, pemetrexed and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Known active Hepatitis B or Hepatitis C
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Phase 1 (safety run-in) | One cycle i.e. 3 weeks
  Dose Limiting Toxicity graded per Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Phase 2 (efficacy) | From date of randomization until date of death from any cause, withdrawal of consent or loss to follow up whichever came first, assessed for up to 35 cycles (2 years)
  Objective Response Rate (ORR) evaluated by RECIST 1.1 and defined as the rate of complete response (CR) + partial response (PR)

SECONDARY OUTCOMES:
ORR | From date of randomization until date of death from any cause, withdrawal of consent or loss to follow up whichever came first, assessed for up to 35 cycles (2 years)
  by baseline PD-L1 expression

CONTACTS AND LOCATIONS:
Overall Officials: James Spicer, MD Prof, Principal Investigator — Guy's Hospital
Locations (13):
- Germany (2):
  - Thoraxklinik Heidelberg gGmbH, Heidelberg, Community of Heidelberg
  - PIUS Hospital Oldenburg, Oldenburg
- Stichting Het Nederlands Kanker Instituut, Amsterdam, Community of Amsterdam, Netherlands
- Spain (9):
  - Servicio de Oncología-El médico del Virgen de la Victoria, Málaga, Andalusia
  - Insituto Oncologico Dr Rosell. Hospital Universitario Quiron Dexeus, Barcelona, Catalonia
  - Hospital Universitario de Vall d'Hebron, Barcelona, Catalonia
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Catalonia
  - Hospital Clinico Universitario de València, Valencia, Horta de València
  - Hospital Universitario 12 Octubre, Madrid, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Puerta del Hierro Majadahonda, Madrid, Madrid
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All unpublished information relating to this trial and/or to the trial treatments is considered confidential by the Sponsor and shall remain the sole property of the Sponsor.
  The Investigator must accept that the Sponsor may use the information from this clinical trial in connection with the development of the IO102, and therefore, may disclose it as required to other Investigators, to government licensing authorities, to regulatory agencies of other governments, stock exchange market, and commercial partners.

REFERENCES:
- [Background] Langer CJ, Gadgeel SM, Borghaei H, Papadimitrakopoulou VA, Patnaik A, Powell SF, Gentzler RD, Martins RG, Stevenson JP, Jalal SI, Panwalkar A, Yang JC, Gubens M, Sequist LV, Awad MM, Fiore J, Ge Y, Raftopoulos H, Gandhi L; KEYNOTE-021 investigators. Carboplatin and pemetrexed with or without pembrolizumab for advanced, non-squamous non-small-cell lung cancer: a randomised, phase 2 cohort of the open-label KEYNOTE-021 study. Lancet Oncol. 2016 Nov;17(11):1497-1508. doi: 10.1016/S1470-2045(16)30498-3. Epub 2016 Oct 10. PMID 27745820
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Iversen TZ, Engell-Noerregaard L, Ellebaek E, Andersen R, Larsen SK, Bjoern J, Zeyher C, Gouttefangeas C, Thomsen BM, Holm B, Thor Straten P, Mellemgaard A, Andersen MH, Svane IM. Long-lasting disease stabilization in the absence of toxicity in metastatic lung cancer patients vaccinated with an epitope derived from indoleamine 2,3 dioxygenase. Clin Cancer Res. 2014 Jan 1;20(1):221-32. doi: 10.1158/1078-0432.CCR-13-1560. Epub 2013 Nov 11. PMID 24218513
- [Background] Andersen MH. Immune Regulation by Self-Recognition: Novel Possibilities for Anticancer Immunotherapy. J Natl Cancer Inst. 2015 Jun 10;107(9):djv154. doi: 10.1093/jnci/djv154. Print 2015 Sep. PMID 26063792